CLINICAL TRIAL: NCT02079389
Title: The Value of Laparoscopic Ultrasound in Patients Undergoing Laparoscopic Resection for Cancer of the Colon or Rectum: A Prospective Randomized Trial
Brief Title: The Value of Laparoscopic Ultrasound in Patients Undergoing Laparoscopic Resection for Cancer of the Colon or Rectum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Svendborg Hospital (Other); Sygehus Lillebaelt (Other); Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, MD Signe Bremholm Rasmussen, MD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20110135
Record Dates: First submitted 2014-02-10; First posted 2014-03-05 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2013-05

CONDITIONS: Colon Cancer; Rectum Cancer; Liver Metastases
Keywords: colon cancer; rectum cancer; laparoscopic ultrasound; LUS; Contrast enhanced ultrasound; CEUS; Peroperative TNM staging; screening for liver metastases
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lap+Lus (Active Comparator): The included patients randomly assigned either to the department's standard laparoscopic (Lap) surgery or standard laparoscopic surgery (lap) plus a LUS examination.
  In the intervention arm the intra-abdominal conditions are also assessed by laparoscopy, but then supplemented with a LUS examination of the primary tumor, liver and retroperitoneum.
  All the included patients are getting a CT scan of the abdomen after 3 months.
  Interventions: Device: Lap+Lus
- laparoscopic examination (Lap) (No Intervention): The included patients randomly assigned either to the department's standard laparoscopic (Lap) surgery or standard laparoscopic surgery (lap) plus a LUS examination.
  In the standard arm (Lap) the conditions at the abdomen is only assessed by laparoscopy immediately prior to the resection.
  All the included patients are getting a CT scan of the abdomen after 3 months.

INTERVENTIONS:
Device: Lap+Lus — In the standard arm (Lap) the conditions at the abdomen is only assessed by laparoscopy immediately prior to the resection. In the intervention arm the intra-abdominal conditions are also assessed by laparoscopy, but then supplemented with a laparoscopic ultrasound examination of the primary tumor, liver and retroperitoneum.
  All patients are given an CT scan of the abdomen after 3 months.
  Other Names: BK medicals; ultrasound solutions
  Arms: Lap+Lus

SUMMARY:
The following project deals with a Danish multicenter trial that evaluates the value of Laparoscopic Ultrasound examination (LUS) in laparoscopic surgery for colon and rectum cancer (CRC).

The project "The value of laparoscopic ultrasound in patients undergoing laparoscopic resection for colon and rectum cancer. - A prospective randomized trial" is part of a ph.d- study at the University of Southern Denmark in collaboration with several surgical departments at hospitals in Southern Denmark.

The primary purpose is to investigate whether the use of laparoscopic ultrasound examination (LUS) will change the stage of the tumor, lymph node and metastasis (TNM stage) and the surgical approach in patients undergoing laparoscopic surgery for colorectal cancer (CRC).

As a secondary objective; an evaluation of the use of LUS will change the treatment strategy for the individual patient with CRC.

As an other objective we wants to investigate whether the use of contrast enhanced ultrasound examination in connection with LUS procedure increases the number of detected liver metastases.

DETAILED DESCRIPTION:
Laparoscopic surgery for cancer in the colon or rectum seems to be equal standing to open surgery with regards to the morbidity, mortality and the oncologic results (radicality and re-lapse frequency and long-term survival). Laparoscopic surgery for colon and rectum cancer is now a well-understood and well-established surgical method, but there are only few randomized trials dealing with the long-term results. The latest inventory work calls for better documentation of long-term results and calls for further randomized studies. Despite this, the number of laparoscopic operations for colorectal cancer (CRC) in Denmark is increasing, and laparoscopic surgery has partially become established as standard treatment for CRC.

Liver metastases are frequent in patients with CRC and about 15-20% of patients already have metastases at the diagnosis. Ultrasound examination during open surgery (IOUS) has shown to be an important diagnostic tool with high sensitivity (98%) and positive predictive value (86%) for detection liver metastases that are undiagnosed on preoperative computed tomography scan (CT) or Positron emission tomography-computed tomography scan (PET-CT). IOUS is considered as the gold standard for hepatic metastases within open surgery for CRC. In laparoscopic surgery this option disappears, but it is likely that Laparoscopic Ultrasound examination (LUS), may provide the same information as found by IOUS.

While laparoscopy and laparoscopic ultrasound examination (LUS) is well established in the staging and treatment of upper gastrointestinal cancers, this method is only sparsely evaluated in the treatment of CRC. There are only very few and older data dealing with the use of LUS in the Tumor - lymph Node and Metastases (TNM) staging in patients with cancer in the colon and rectum. Several small studies have investigated the use of LUS to evaluate the M-stage in laparoscopic colorectal surgery and all studies show an increased detection of liver metastases. Overall, seems LUS to be better than the current pre-operative image modalities, and the LUS and the IOUS has also been found to be able to locate small tumors in the colon.

Based on the above, a recent review concluded that the data about the routine use of laparoscopy and LUS in patients with CRC are not sufficient, but that LUS probably could be used for assessment of the liver, liver-metastases and non-regional lymph nodes. There are no randomized studies dealing with the use of LUS in laparoscopic surgery for CRC.

It is not a standard routine to use LUS of the liver, tumor and retroperitoneum during laparoscopic surgery for CRC.

In prospective and blinded studies a percutaneous contrast-enhanced ultrasound examination (CEUS) of the liver proved to be able to detect significantly more liver metastases from CRC than conventional percutaneous ultrasound.

With the new second-generation contrast agents CEUS seems to be equivalent to the contrast-enhanced CT and Magnetic resonance imaging (MRI) for detection liver-metastases.

Liver metastases are frequent in patients with CRC and the use of intraoperative ultrasound (IOUS) during open surgery for CRC, has previously been regarded as the gold standard. Contrast-enhanced IOUS (CE-IOUS) during open surgery for CRC is only sparsely evaluated, but has been shown to increase sensitivity for detection liver-metastases. There is on the other hand, not found literature that has been describing the use of laparoscopic CE-IOUS during laparoscopic surgery for CRC.

With this project we want to elucidate whether the use of LUS in laparoscopic surgery for CRC will alter the patient's TNM stage and surgical approach and whether potential changes have any clinical consequence for the individual patient. Furthermore, we wish to investigate whether contrast-enhanced LUS increases detection rate for liver metastases.

Method The study is designed as a prospective, randomized multicenter study and include 280 patients.

At the Department of Surgery, Odense University Hospital, they annually conducted around 150 laparoscopic resections for CRC, but the department has a selected patient material. To get a representative sample of patients with CRC, and to get included as many patients as possible within the given timeframe, the project will therefore be conducted as a multicenter study.

The participating centers perform all laparoscopic CRC surgery at a high level, and both the technical equipment and the necessary scanning competencies are available on the departments involved.

Prior to the start of the project, the surgeons of the included departments will be trained in the LUS method, so that assessment and description of the intra-abdominal findings are standardized.

They included patients randomly assigned either to the department's standard laparoscopic surgery or standard laparoscopic surgery plus a LUS examination.

In the standard arm the conditions at the abdomen is only assessed by laparoscopy immediately prior to the resection.

In the second group the intra-abdominal conditions are also assessed by laparoscopy, but then supplemented with a LUS examination of the primary tumor, liver and retroperitoneum.

Both laparoscopy and LUS will take place just prior in to the operation itself and will not require further intervention or additional portholes.

If there at the LUS examination is found undiagnosed liver metastases or lymph nodes outside the planned operation field, then the patient is sent to the Department of Surgery A, Odense University Hospital, for a multidisciplinary tumor conference.

In cases where the LUS examination suspects liver metastases and / or remove lymph node metastases in patients who are included in the project at the Department of Surgery A, Odense University Hospital, then a intraoperative LUS-guided fine-needle aspirations- biopsy (FNA) or tru-cut biopsy will be performed and marked with a little silver pin. The latter is used for follow-up after pretreatment and to locate potential rest tumor.

All other patients follow the Departments usual routines for adjuvant therapy.

Those patients who are selected for laparoscopic resection at the Department A, University Hospital also offers to participate in a contrast-enhanced laparoscopic Ultrasound examination during surgery. A specialist with skills in contrast-enhanced ultrasound will perform the examination.

Before the contrast study is performed the surgeon notes the findings after conventional LUS, so that the patients examined at University Hospital also is part of the total material on an equal footing with those scanned in the other departments.

All patients included in the project will undergo a three-phase control computed tomography (CT) scan 3 months after surgery. This is to evaluate whether there might be overlooked metastases in the laparoscopy and LUS evaluation.

All the information about the patients are entered and recorded in a database. Information on death will be deducted from the Civil Registration and local administrative databases.

After completion of the inclusion of patients, the two arms will be compared with account of changes in the TNM-stage and surgical approach in relation to the pre-operative assessment.

The possible changes are evaluated from strict, predefined criteria and are assessed whatever they have clinical relevancy, and finally the potential effect of contrast-enhanced LUS compared to LUS alone is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with colon and rectum cancer without known metastasis
* Patients who gives informed consent
* Patients who are referral to laparoscopic surgery

Exclusion Criteria:

* Patients who are not able to give informed consent
* Patients who are under 18 of age Patients with known metastasis.
* Patients who are allergic to contrast agents
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
A change in the stage of Tumor, lymph Node and metastases (TNM-stage) | 3 months
  When using laparoscopic ultrasound examination (LUS) during laparoscopic resection for colon and rectum cancer, it is possible to scan the tumor, lymph nodes around the tumor, retroperitoneum and the liver. Thereby it is possible to make a preoperative TNM staging. Will the use of LUS change the stage of Tumor lymph Node and Metastases (TNM stage) compared to the preoperative TNM evaluation. The procedure LUS takes approximately 5 to 10 minutes. Tree months after surgery the patients will get a CT scan of the liver to ensure that the LUS did not miss any metastasis.

SECONDARY OUTCOMES:
A change in the postoperative treatment strategy | 3 months
  Will the use of laparoscopic ultrasound (LUS) during laparoscopic resection for colon and rectum cancer make af change in the patients treatment strategy. While using LUS during laparoscopic resection for colon and rectum cancer the tumor, lymph nodes, retroperitoneum and the liver is scanned with ultrasound and a peroperative TNM staging are done. If there are any differences in the peroperative TNM stage compared to the preoperative TNM stage, will it then have a consequence for the patient. For example: It could be a biopsy from a potential metastasis or enlarged lymph node ect. Will the changes alter the primary treatment strategy for the patient.

OTHER OUTCOMES:
Does the use of contrast enhanced ultrasound examination during surgery for colon and rectum cancer provides more findings of liver metastases? | 10 minutes
  The patients who are undergoing laparoscopic colon and rectum cancer surgery at the surgical department Odense University Hospital will get a contrast enhanced laparoscopic ultrasound examination.The laparoscopic ultrasound examination (LUS) is done at first. Then it will be supplied with a contrast enhanced examination done by a specialist in liver surgery. The liver is the primary focus and there is only searched for liver metastases. The examination will take about 10 minutes. If there is found a liver metastasis or if any are suspected the specialist i liver surgery will make sure that the patient will get the right treatment for the metastasis.

CONTACTS AND LOCATIONS:
Overall Officials: Signe bremholm Rasmussen, MD, Study Director — Odense University Hospital; Michael Bau Mortensen, professor, Principal Investigator — Odense University Hospital; Claus Fristrup, ph.d, Principal Investigator — Odense University Hospital
Locations (4):
- Denmark (4):
  - Esbjerg Hospital, Esbjerg, Esbjerg
  - Odense University Hospital, Odense, Odense
  - Svendborg Hospital, Svendborg, Svendborg
  - Lillebaelt Hospital, Vejle, Vejle

REFERENCES:
- [Derived] Ellebaek SB, Fristrup CW, Hovendal C, Qvist N, Bundgaard L, Salomon S, Stovring J, Mortensen MB. Randomized clinical trial of laparoscopic ultrasonography before laparoscopic colorectal cancer resection. Br J Surg. 2017 Oct;104(11):1462-1469. doi: 10.1002/bjs.10636. PMID 28895143